CLINICAL TRIAL: NCT06977100
Title: Examining the Feasibility and Acceptability of a Journaling Intervention in Alleviating Temporomandibular Pain
Brief Title: Journaling Intervention for Temporomandibular Disorder (TMD) and Chronic Overlapping Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB202500344
Record Dates: First submitted 2025-05-08; First posted 2025-05-18 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-05

CONDITIONS: Temporomandibular Disorders (TMD)
Keywords: Temporomandibular Disorder; Gratitude Journaling; Resilience; Pain Intensity; Pain Interference; Chronic Pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Pain; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gratitude Intervention (Experimental)
  Interventions: Behavioral: Gratitude
- General Wellness (Active Comparator)
  Interventions: Other: General Wellness

INTERVENTIONS:
Behavioral: Gratitude — Participants in this group will receive a gratitude journal where they will be asked to write down three things they are grateful for each day and reflect why they are grateful for these things. Journaling will take place from the comfort of their home on three days of their choice per week, for a total duration of two weeks.
  Arms: Gratitude Intervention
Other: General Wellness — Participants in this group will receive a general wellness journal where they will be asked to reflect on three things that happened, or they did during the day (daily activities). Journaling will take place from the comfort of their home on three days of their choice per week, for a total duration of two weeks.
  Arms: General Wellness

SUMMARY:
The goal of this clinical trial is to learn whether a 2-week gratitude journaling activity is feasible and acceptable for individuals with Temporomandibular Disorder (TMD) and chronic overlapping pain. The study will also look at whether this activity is helpful in reducing pain and how much it interferes with daily life.

The primary aims of this study are to:

* Assess whether individuals with TMD and chronic overlapping pain are able to complete the 2-week gratitude journaling activity as planned (feasibility).
* Evaluate how acceptable participants find the gratitude journaling activity (acceptability).

The secondary aim of this study is to:

• Explore whether the gratitude journaling activity reduces pain and its impact on daily life, compared to a general wellness journaling activity.

Participants will:

* Attend two in-person visits to complete questionnaires and take part in tests that measure how sensitive they are to pressure and heat.
* Complete a 2-week journaling activity at home, writing in their journal on three days of their choice per week.

ELIGIBILITY:
Inclusion Criteria:

* participants between the ages of 18 and 80
* pain in the temporomandibular (TMD) region (jaw and/or temple area)
* duration of pain is at least 3 months
* average pain score ≥4 on a 0-10 numerical rating scale over the past week
* have at least one additional chronic overlapping pain condition (COPC) including fibromyalgia, irritable bowel syndrome, migraine-type headache, tension-type headache, low back pain, interstitial cystitis/painful bladder syndrome or chronic prostatitis, myalgic encephalomyelitis/chronic fatigue syndrome, vulvodynia, and painful endometriosis.
* able to read, understand, and write in English.

Exclusion Criteria:

* history of TMD surgery
* neoplasm or injury/trauma to the TMD area
* cancer-related pain
* scheduled for any surgeries during the study time-frame
* current participation in another clinical trial or psychological treatment for any pain-related condition that would interfere with study outcomes
* pregnant or lactating
* severe motor impairments (e.g., muscular dystrophy)
* severe psychiatric conditions (e.g., uncontrolled mood disorders)
* severe neurological or cognitive impairments (e.g., uncontrolled Parkinson's disease)
* any other conditions that in the opinion of study investigators could make participation in the study unsafe
* use of opioids within 48 hours prior to laboratory visit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Participant Retention | Baseline to Week 4
  Percentage of participants who initiate treatment/intervention and complete the post-intervention assessment at the 4-week time-point.
Treatment Satisfaction | Week 4
  Single-item Treatment Satisfaction Questionnaire: Response to self-reported item assessing overall satisfaction with the treatment. The item is rated on a 1 to 4 scale (1 = Quite Dissatisfied to 4 = Very Satisfied) with the mean value calculated. A higher score indicates greater satisfaction with the treatment.

SECONDARY OUTCOMES:
Pain Intensity | Baseline, Week 4
  The PROMIS-Pain Intensity short form is a 3-item measure assessing pain intensity over the past 7 days (i.e., "how intense was your pain at its worst"), as well as current level of pain. The total score for the PROMIS Pain Intensity short form will be calculated by summing the numerical values of the responses to each of the three items. After obtaining the total raw score, it will then be converted into a T-score, which standardizes the score with a mean of 50 and a standard deviation of 10, based on the general U.S. population.
Pain Interference | Baseline, Week 4
  The PROMIS-Pain Interference short form is an 8-item measure assessing the extent to which pain interferes with physical, mental, cognitive, emotional, recreational and social activities over the past 7 days (i.e., "how much did pain interfere with work around home"). The total score for the PROMIS-Pain Interference short form will be calculated by summing the numerical values of the responses to each of the eight items. After obtaining the total raw score, it will then be converted into a T-score, which standardizes the score with a mean of 50 and a standard deviation of 10, based on the general U.S. population.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No